CLINICAL TRIAL: NCT03703947
Title: Study of Biomarker Profiling to Unravel the Intertwined Pathophysiology of Coronary Artery Disease and Abdominal Aortic Aneurysm
Brief Title: Biomarker Profiling in Abdominal Aortic Aneurysm Patients
Acronym: BIOMArCS-AAA
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Maasstad Hospital (Other)
Responsible Party: Principal Investigator, Isabella Kardys, Principal investigator, associate professor, Erasmus Medical Center
Other Study IDs: MEC-2017-019
Record Dates: First submitted 2018-10-08; First posted 2018-10-12 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal Aortic Aneurysm; Biomarkers
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (EDTA plasma, citrate plasma, serum, DNA) is taken at the day of inclusion and at follow-up visits, which will be performed every 6 months, until the end of the 2-years scheduled follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Watchful-waiting group: The prospective, longitudinal part of the study will include an arm with 120 AAA watchful waiting patients, with a 24-month follow-up period. Clinical data collection, and blood sampling will be conducted at baseline, and at 6, 12, 18 and 24 months for all patients. CT will be conducted at baseline and 12 and 24 months. Quality of life and depression questionnaires will be performed at baseline, at 12 and 24 months of follow-up in all patients.
- EVAR group: The prospective, longitudinal part of the study will include an arm with 120 AAA patients undergoing endovascular aneurysm repair (EVAR), with a 24-month follow-up period. Clinical data collection, and blood sampling will be conducted at baseline, at 1 month after EVAR and at 6, 12, 18 and 24 months after EVAR. CT will be conducted at baseline, at 1 month after EVAR and at 12 and 24 months after EVAR patients. Quality of life and depression questionnaires will be performed at baseline, at 1 month, at 12 and 24 months of follow-up after EVAR.
- Cross-sectional group (after EVAR): A cross-sectional study will be performed in 200 patients treated for AAA with EVAR in the past years. In these patients, clinical data collection, blood sampling, ultrasound and CT will be performed at their next regular outpatient clinic visit.

SUMMARY:
The BIOMArCS-AAA study aims to investigate the associations of (temporal patterns of) blood biomarkers with aneurysm growth in patients with abdominal aortic aneurysm (AAA), with particular attention to biomarkers that have demonstrated prognostic value for adverse disease outcomes in coronary artery disease and biomarkers for the main genetic pathways associated with AAA.

DETAILED DESCRIPTION:
BIOMArCS-AAA is an observational, multicenter study. Patients with an abdominal aortic aneurysm (AAA) will be recruited through the vascular surgery outpatient clinic of Erasmus MC and Maasstad Ziekenhuis, the Netherlands. The prospective, longitudinal part of the study will include an arm with 120 AAA watchful waiting patients and an arm with 120 AAA patients undergoing endovascular aneurysm repair (EVAR), both with a 24-month follow-up period. Clinical data collection, and blood sampling will be conducted at baseline, at 1 month after EVAR and at 6, 12, 18 and 24 months for all patients. CT will be conducted at baseline and 12 and 24 months, plus at 1 month in the EVAR patients. Quality of life and depression questionnaires will be performed at baseline, at 12 and 24 months of follow-up in all patients, and at 1 month only in EVAR patients. Additionally, a cross-sectional study will be performed in 200 patients treated for AAA with EVAR in the past years. In these patients, clinical data collection, blood sampling, ultrasound and CT will be performed at their next regular outpatient clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Capable of understanding and signing informed consent AND one of the following

  1. Diagnosis of AAA, with a diameter ≥40mm, based on any imaging technique and treated by watchful waiting strategy (Prospective longitudinal study, Arm 1 watchful waiting group)
  2. Planned to undergo EVAR for AAA (Prospective longitudinal study, Arm 2 EVAR group)
  3. Underwent EVAR for AAA in past years (Cross-sectional study)

Exclusion Criteria:

* Patients with isolated iliac artery aneurysm, traumatic aneurysm, anastomotic aneurysm and infectious aneurysm
* Patients with a clinical diagnosed thoracic aneurysm (i.e. located in the chest, above the diaphragm)
* Coexistent condition with life expectancy ≤ 1 year
* Dialysis dependent, (end stage) renal disease patients
* Women of childbearing age
* Linguistic barrier
* Unlikely to appear at all scheduled follow-up visits

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with an abdominal aortic aneurysm, visiting the outpatient clinic.
Sampling Method: Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2017-03-23 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Volume of the aneurysm sac | Measured cross-sectionally, as well as repeatedly in the longitudinal part of the study by CT scan imaging during 24 months of follow-up.
  The primary study endpoint is volume of the aneurysm sac. This will be measured cross-sectionally, as well as repeatedly in the longitudinal part of the study by CT scan imaging during 24 months of follow-up.

SECONDARY OUTCOMES:
Maximal diameter of the aneurysm | Measured cross-sectionally, as well as repeatedly in the longitudinal part of the study during 24 months of follow-up.
  Maximal diameter of the aneurysm by CT scan imaging
Number of deceased patients due to all-cause mortality | During 24 months of follow-up in the longitudinal part of the study.
  All-cause mortality
Number of AAA-related adverse events in watchful waiting group | During 24 months of follow-up in the watchful-waiting patients of the longitudinal part of the study.
  AAA related death, AAA rupture, or any AAA-related intervention.
Number of AAA-related adverse events in EVAR patients | During 24 months of follow-up in the EVAR patients of the longitudinal part of the study.
  Endoleaks, migration >10 mm, device integrity failure, AAA-related death, late postimplantation AAA rupture, or any AAA-related secondary intervention.
Number of patients with cardiovascular events | Cross-sectionally and during 24 months of follow-up in the longitudinal part of the study.
  Cardiovascular events: i.e. cardiovascular death, myocardial infarction, percutaneous coronary intervention (PCI), coronary artery bypass grafting (CABG).
Quality of life measured according to the EuroQol questionnaire | Measured repeatedly during 24 months of follow-up in the longitudinal part of the study.
  The validated questionnaire EuroQol will be used to assess health related quality of life
Depression measured according to the Hospital Anxiety and Depression Scale questionnaire | Measured repeatedly during 24 months of follow-up in the longitudinal part of the study.
  The Hospital Anxiety and Depression Scale (HADS) will be assessed to adjust for depression and anxiety in combination with the 2-item Patient Health Questionnaire (PHQ-2).

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Kardys, MD, PhD, Study Chair — Erasmus Medical Center; Eric Boersma, MSc, PhD, Study Director — Erasmus Medical Center; Hence JM Verhagen, MD, PhD, Principal Investigator — Erasmus Medical Center; Bram Fioole, MD, PhD, Principal Investigator — Maasstad Hospital
Locations (2):
- Netherlands (2):
  - Erasmus Medical Center, Rotterdam, South Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vanmaele A, Bouwens E, Hoeks SE, Kindt A, Lamont L, Fioole B, Budde RP, Ten Raa S, Hussain B, Oliveira-Pinto J, Ijpma AS, van Lier F, Akkerhuis KM, Majoor-Krakauer DF, de Bruin JL, Hankemeier T, de Rijke Y, Verhagen HJ, Boersma E, Kardys I. Targeted plasma multi-omics propose glutathione, glycine and serine as biomarkers for abdominal aortic aneurysm growth on serial CT scanning. Atherosclerosis. 2024 Nov;398:118620. doi: 10.1016/j.atherosclerosis.2024.118620. Epub 2024 Oct 2. PMID 39378678
- [Derived] Bouwens E, Vanmaele A, Hoeks SE, Verhagen HJ, Fioole B, Moelker A, Ten Raa S, Hussain B, Oliveira-Pinto J, Bastos Goncalves F, Ijpma AS, Hoefer IE, van Lier F, Akkerhuis KM, Majoor-Krakauer DF, Boersma E, Kardys I. Circulating biomarkers of cardiovascular disease are related to aneurysm volume in abdominal aortic aneurysm. Vasc Med. 2023 Oct;28(5):433-442. doi: 10.1177/1358863X231181159. Epub 2023 Jul 3. PMID 37395286